CLINICAL TRIAL: NCT05111340
Title: Securing the Immediate Perioperative Walk: Creating and Validating a Score.
Acronym: Déambu
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ramsay Générale de Santé (Other)
Collaborators: European Clinical Trial Experts Network (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 2017-A02478-45
Record Dates: First submitted 2021-10-27; First posted 2021-11-08 (Actual); Last update posted 2021-11-08 (Actual); Status verified 2021-10

CONDITIONS: Wandering Behavior; Anesthesia
MeSH Terms: conditions — Wandering Behavior

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Adult patients undergoing sedation with or without associated local anesthesia (Experimental)
  Interventions: Behavioral: Perioperative score

INTERVENTIONS:
Behavioral: Perioperative score — Creation and validation of a perioperative walk score. The patient has to answer different items.

SUMMARY:
The aim of this study is to set up a pre and postoperative ambulation score on a population of adult patients and undergoing outpatient surgery operated under locoregional anesthesia and sedation.

ELIGIBILITY:
Inclusion Criteria:

* Patient over 18 years-old
* Patient undergoing sedation with or without associated local anesthesia
* Patient having giver their consent
* Patient are benefiting from a social protection insurance
* Patient hospitalized as part of the outpatient for ophthalmologic surgery or upper limb surgery, plastic surgery or surgery for implantation of a vascular access device

Exclusion Criteria:

* Patient whose surgery is performed on the lower limbs
* Patient with psychiatric disorders
* Patient with dementia
* Patient who has already participated in this same study (ex: cataract the second eye is made a few weeks after the first)
* Patient's refusal to participate in the study
* Protected patients: Adults under guardianship, curatorship or other legal protection, deprived of their liberty by judicial or administrative decision; Pregnant, breastfeeding or parturient woman; Hospitalized without consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 525 (Actual)
Dates: Start 2018-04-23 (Actual); Primary Completion 2021-05-01 (Actual); Study Completion 2021-06-12 (Actual)

PRIMARY OUTCOMES:
The validity of the perioperative walk score | 1 day
  The validity of the score will be assessed using the theory of item response (TRI). This theory is based on the correlations between the items of the score.

CONTACTS AND LOCATIONS:
Locations (1):
- Hôpital privé Arras les Bonnettes, Arras, France